



St George's Hospital Blackshaw Road London SW17 0QT

Direct Line: 020 8672 1255 Direct Fax: 020 8672 5304

www.st-georges.org.uk

IRAS ID: 284337

Centre Number: St George's University of London

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: Can MRI-based computational modelling of the heart be used to predict critical substrate in scar-dependent ventricular tachycardia ablation?

Name of Researchers: Dr Michael Waight, Dr Anthony Li, Dr Magdi Saba, Cardiovascular Sciences Department, St George's University of London, Cranmer Terrace, SW17 0RE

| Р | lease | ın | ıtıa | ı | hox |
|---|-------|----|------|---|-----|

| Plea | se initial box | | |
|---|---|---|---|
| 1. | | d 12/02/2021 (version 1.1) for the he information, ask questions and | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from St George's University of London, St George's Hospital NHS Foundation Trust or from regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| 4. | I agree that data from my cardiac MRI will be shared with Johns Hopkins University, USA as described in the Patient Information Sheet. | | |
| 5. | . I agree to take part in the above study. | | |
| 6. | i. I agree to my GP being informed of my involvement. | | |
| ——<br>Nam | e of participant | <br>Date | Signature |
| Name of person taking consent | | Date | Signature |